CLINICAL TRIAL: NCT03546647
Title: Toric Contact Lens Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Kathryn Richdale, Associate Professor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Study00000682
Record Dates: First submitted 2018-05-18; First posted 2018-06-06 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Toric, Then Sphere (Experimental): Participants who received Toric contact lenses first and spherical lenses after 10 days
  Interventions: Device: Dailies Aqua Comfort Plus Toric; Device: Dailies Aqua Comfort Plus Sphere
- Sphere, Then Toric (Experimental): Participants who received Spherical contact lenses first and Toric lenses after 10 days
  Interventions: Device: Dailies Aqua Comfort Plus Toric; Device: Dailies Aqua Comfort Plus Sphere

INTERVENTIONS:
Device: Dailies Aqua Comfort Plus Toric — Daily disposable soft toric contact lens
Device: Dailies Aqua Comfort Plus Sphere — Daily disposable soft spherical contact lens

SUMMARY:
This study seeks to quantify digital visual performance and subjective visual acceptance of toric contact lenses as compared to spherical lenses in low to moderate astigmatic patients.

DETAILED DESCRIPTION:
This is a prospective, single site, randomized, masked, crossover study. This study will evaluate the ability of toric contact lenses to decrease signs and symptoms of asthenopia and improve digital reading performance. Symptoms and objective near vision outcomes will be measured at baseline and after 1 week of wear with each correction.

ELIGIBILITY:
Inclusion

+6.00 to -6.00 D vertexed sphere power and -0.75 to -1.50 D vertexed refractive cylinder in the right and left eyes Best corrected acuity of 20/25 or better in each eye Self report of at least 4 hrs/day using digital devices Current/established soft contact lens wearer (has worn contact lenses in the past year)

Exclusion An optometrist or optometry student History of ocular pathology or surgery Binocular vision disorder (i.e., tropia, convergence or accommodative insufficiency) Gas permeable lens wear for at least 3 months Presbyopic (based on refraction)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Richdale, OD, PhD, Principal Investigator — University of Houston College of Optometry
Locations (1):
- University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 participants were screened for eligibility between March and November 2018.
Pre-assignment Details: 35 of 37 participants were randomized. Of those not randomized, 2 did not meet inclusion criteria. One randomized subject was removed from the study due to an adverse event.
Groups:
- Sphere, Then Toric: Participants who received Sphere contact lenses first and Toric lenses after 10 days
Period: Overall Study
Arm/Group | Toric, Then Sphere | Sphere, Then Toric
Started | 18 | 17 (34)
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Toric group:
  Participants who received Toric contact lenses first and spherical lenses after 10 days
  Sphere group:
  Participants who received spherical contact lenses first and Toric lenses after 10 days
Arm/Group | All Study Participants
Number analyzed (Participants) | 34
Age, Customized [Mean (Standard Deviation); unit: years]
  Male | 22.2 (2.7)
  Female | 27.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Near Visual LogMAR Acuity
Description: High contrast LogMAR visual acuity was assessed at 40 cm using the M&S Clinical Trial Suite system (Niles, Illinois, USA). The system was calibrated according to the manufacturer's directions every day, prior to use. Testing was performed binocularly. The test started at 20/200 and continued until three letters were missed on a line.
Time Frame: 10 +/- 2 days
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Toric: Participants who wore Toric contact lenses for 10 days
- Sphere: Participants who wore Spherical contact lenses for 10 days
Arm/Group | Toric | Sphere
Number analyzed (Participants) | 34 | 34
LogMAR | -0.09 (0.07) | -0.02 (0.09)

ADVERSE EVENTS:
Time Frame: 10 ± 2 days for each intervention
Description: AE information was collected at each study visit
Groups:
- Toric: Soft toric contact lens
  Dailies Aqua Comfort Plus Toric: Daily disposable soft toric contact lens
- Sphere: Soft sphere contact lens
  Dailies Aqua Comfort Plus Sphere: Daily disposable soft spherical contact lens
Arm/Group | Toric | Sphere
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 1/34 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric (N=34) | Sphere (N=34)
Keratitis (Eye disorders) | 1 (1) | 0 (0) — superficial punctate keratitis > grade 2 OU

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03546647/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03546647/SAP_001.pdf